CLINICAL TRIAL: NCT00510029
Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of GAP-134 Administered Intravenously as a 24-Hour Infusion to Healthy Subjects.
Brief Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of GAP-134 Administered Intravenously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: 3205K2-1000
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — 1-(2-aminoacetyl)-4-benzamidopyrrolidine-2-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- GAP-134, IV and Oral (Other): Experimental; Active Comparator; Placebo
  Interventions: Drug: GAP-134

INTERVENTIONS:
Drug: GAP-134 — atrial fibrillation 24-hr IV infusion; 1-minute IV bolus; PO

SUMMARY:
The study will assess the safety, tolerability and pharmacokinetics of single intravenous (IV) doses of GAP-134 in healthy subjects. GAP-134 will be administered as a 24-hour infusion.

ELIGIBILITY:
Inclusion Criteria

* Generally healthy men and women of nonchildbearing potential (WONCBP), aged 18 to 50 years.
* Body Mass Index (BMI) range of 18 to 30 kg/m2.
* Blood serum creatinine levels less than or equal to the upper limit of normal.

Exclusion Criteria

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any history of clinically important cardiac arrhythmias and familial history of long QT syndrome or unexpected cardiac death.
* History of drug and alcohol abuse, positive HIV, HCV, and/or HBs Ag test, and any clinically important deviation from normal limits in physical examination, vital signs, 12-lead ECGs, or clinical laboratory test results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single ascending IV doses of GAP-134 administered as 24-hour continuous infusions and as single bolus injection of GAP-134 in healthy subjects | 3-4 months

SECONDARY OUTCOMES:
To provide the initial Pharmacokinetic (PK) profile of single ascending IV doses (24 hour and 1-minute) and the initial PK assessment of the bioavailability of an oral formulation of GAP-134 under fasting conditions in healthy subjects | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States